CLINICAL TRIAL: NCT03699202
Title: A Randomised, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety and Tolerability of Orally Administered AK0529 in Adults With Respiratory Syncytial Virus Infection
Brief Title: Anti-RSV Study in Chinese Patients (ASCENT)
Acronym: ASCENT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Ark Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AK0529-2002
Record Dates: First submitted 2018-10-05; First posted 2018-10-09 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: RSV,AK0529,Chinese
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — ziresovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 100mg AK0529 Arm (Experimental): Patients randomised into this arm will be orally administered with 100mg AK0529 q.d. for five days.
  Interventions: Drug: AK0529
- 200mg AK0529 Arm (Experimental): Patients randomised into this arm will be orally administered with 200mg AK0529 q.d. for five days.
  Interventions: Drug: AK0529
- 300mg AK0529 Arm (Experimental): Patients randomised into this arm will be orally administered with 300mg AK0529 q.d. for five days.
  Interventions: Drug: AK0529
- Placebo Arm (Placebo Comparator): Patients randomised into this arm will be orally administered with placebo q.d. for five days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AK0529 — AK0529 is a novel compound being developed for the treatment of RSV infection. The capsule containing enteric coated AK0529 pellets will be orally administered to patients at one of a 100mg, 200mg or 300mg dose level.
  Other Names: Ziresovir
  Arms: 100mg AK0529 Arm; 200mg AK0529 Arm; 300mg AK0529 Arm
Drug: Placebo — The placebo is made with the same smell and appearance as AK0529 but without the active ingredients. The placebo supplements are composed of microcrystaline cellulose pellet.
  Arms: Placebo Arm

SUMMARY:
This is a randomised, double-blind, placebo-controlled, multicentre, phase 2 study to evaluate the efficacy, safety and tolerability of orally administered AK0529 in Chinese adults with RSV infection.

DETAILED DESCRIPTION:
This is a randomised, double-blind, placebo-controlled, multicentre, phase 2 study in Chinese adult outpatients with RSV infection. Approximately 160 eligible patients who have been recently diagnosed with RSV infection are planned to be enrolled into the study. Symptom scores of patients before and after treatment will be evaluated. Meanwhile, nasopharyngeal samples and blood samples will be collected for virological and pharmacokinetics evaluations. The evaluation of the safety and tolerability will include AE/SAE, vital signs, physical examination, laboratory examination and 12-lead ECGs. The total study duration for each patient will be 20 days.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 75 years, inclusive.
* Confirmed with RSV infection by rapid diagnostic testing.
* New onset with documentation of the following symptoms within 72 hours prior to the start of screening: Respiratory symptoms: runny nose, stuffy nose, sneezing, sore throat, earache, cough, shortness of breath; Systemic symptoms: headache, fatigue / lethargy, fever, and muscle and / or joint ache. The patient must have four symptoms of above, and at least one of these must be respiratory symptom in nature.
* Able and willing to provide written informed consent and to comply with the study protocol.

Exclusion Criteria:

* The patient has taken, is taking or needs to take any antiviral medication (e.g. ribavirin, Chinese medicine or herbs with effects of treating respiratory tract infection) within the 72 hours prior to screening.
* Awareness of concomitant infections of respiratory viruses (eg, influenza A, B), bacterial or fungal infections, including systemic bacterial or fungal infections within 7 days prior to screening or during the screening period.
* Patient frailty was evaluated as "Vulnerable" or worse according to the Clinical Frailty Scale with a score ≥ 4 at screening.
* Awareness of having positive results on HBsAg or HCV antibody or HIV (HIV 1 or HIV 2).
* Patient with active tuberculosis or is taking antituberculosis treatment.
* Patient with severe gastrointestinal disease which could impact drug absorption, eg, vomiting, malabsorption syndrome, or short bowel syndrome caused by necrotizing enterocolitis.
* Patient with any congenital heart disease, acute or chronic heart failure, ischemic heart disease, or congenital long QT syndrome, or any clinical manifestation resulting in QT interval prolongation.
* Patient with malignant tumor.
* Patient has received or is waiting for bone marrow, stem cell or solid organ transplantation.
* Patient with any immune-related disease to be treated within 12 months prior to screening.
* Patient with clinical laboratoy test values of ≥ 2x the upper limit of normal (ULN) for alanine aminotransferase or aspartate aminotransferase, or >1x ULN for total bilirubin, or >1.5xULN for serum creatinine.
* Patient with electrolyte disorders, eg, hypokalemia, hypocalcemia, or hypomagnesemia.
* Patient with history of drug or alcohol abuse within 12 months prior to screening ("alcohol abuse" definition is >14 units per week: 1 unit = 10mL Alcohol, or 250mL of 4% beer, or 25 mL of 40% spirit, or 75 mL of 13% wine).
* Patient has allergy or hypersensitivity to study medication or its compositions.
* Female patient with positive pregnancy test result or is lactating.
* Patient with fertility refusing to use medically effective contraceptives during the study or within three months of the end of study.
* Patient participated in an investigational drug or device study within 60 days prior to screening.
* Patient who in the opinion of the investigator, is deemed as ineligible for the study, including patients who are with active psychiatric disease, or are taking psychiatric medication.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2019-03-29 (Actual); Primary Completion 2020-01-31 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of symptom score | From Day 0 to Day 5
  To evaluate the change of patient-reported symptom score in AK0529 arms compared with the change in placebo arm after treatment. The scale is Wang bronchiolitis score and the total score is reported with a range from 0 to 12. A decreasing value of total score represents clinical improvement. Subscales are not applicable in this symptom score.
Incidence of adverse events during the study | From Day -3 to Day 14
  An adverse event (AE) is any untoward medical occurrence in a clinical investigation patient administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Subject withdrawals due to treatment-emergent adverse events | From Day -3 to Day 14
  A treatment-emergent adverse event (TEAE) is an AE that first appears during treatment, which was absent before or which worsens relative to the pre-treatment state.

SECONDARY OUTCOMES:
Area under curve change of viral load | From Day 0 to Day 5
  The antiviral effects in adults with RSV infection are to be determined by measuring the RSV viral load area under the curve from baseline to last administration of study medication .

CONTACTS AND LOCATIONS:
Overall Officials: Ark Clinical Trial, Study Director — info@arkbiosciences.com
Locations (22):
- China (22):
  - Beijing Ditan Hospital, Beijing, Beijing Municipality
  - Beijing Anzhen Hospital, Beijing, Beijing Municipality
  - Quanzhou First Hospital, Quanzhou, Fujian
  - Huizhou Municipal Central Hospital, Huizhou, Guangdong
  - The Second Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Sanya Central Hospital, Sanya, Hainan
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Jiangsu Taizhou People's Hospital, Taizhou, Jiangsu
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - People's Hospital of Deyang City, Deyang, Sichuan
  - Suining Central Hopital, Suining, Sichuan
  - China-Japan Friendship Hospital, Beijing
  - Beijing Pinggu Hospital, Beijing
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu
  - Nantong First People's Hospital, Nantong
  - Shanghai East Hospital, Shanghai
  - Central Hospital of Minhang District, Shanghai, Shanghai
  - Shenzhen People's Hospital, Shenzhen
  - Xiangtan Central Hospital, Xiangtan
  - Xinxiang First People's Hospital, Xinxiang
  - Affiliated Hospital of Zunyi Medical University, Zunyi

IPD SHARING:
Plan to Share IPD: No